CLINICAL TRIAL: NCT04536454
Title: A Phase 1/2, Open-label Study to Assess Safety, Tolerability, Biodistribution, Radiation Dosimetry and PET Imaging Characteristics of [18F]FPyGal in Comparison to in Vitro Diagnostics for the Assessment of Senescence in Oncological Patients
Brief Title: Study to Assess Safety and PET Imaging Characteristics of a Novel Senescence-specific Radiotracer [18F]FPyGal (2-[Fluorine-18]Fluoro-3-pyridinyl-β-D-galactopyranoside)
Acronym: SenPET
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: iFIT-01
Record Dates: First submitted 2020-08-20; First posted 2020-09-02 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2020-08

CONDITIONS: Cancer
Keywords: Senescence; [18F]FPyGal; PET / CT; PET / MRI
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [18F]FPyGal (Experimental): Cancer patients will first be treated with a tumor type-specific neo-adjuvant chemotherapy regimen (standard-of-care); subsequently, they will undergo surgical resection of their primary tumors in a curative intention.
  After the end of the neo-adjuvant therapy a tracer injection with [18F]FPyGal solution will be administered (study intervention). Immediately after the injection a dynamic PET/MR imaging of the tumor sites including heart or large arterial blood pools will be conducted over 90 minutes.
  Interventions: Drug: [18F]FPyGal

INTERVENTIONS:
Drug: [18F]FPyGal — Radiotracer for PET-imaging
  Other Names: non-invasive imaging of tumor senescence

SUMMARY:
It is of particular interest to find out whether it is possible to use the novel radiotracer [18F]FPyGal to be tested to detect areas after standard tumor therapy that contain resistant (therapy-resistant) tumor cells. This resistance phenomenon in tumor tissues, which may be visualized with the radiotracer [18F]FPyGal, is called tumor senescence.

DETAILED DESCRIPTION:
The so-called tumor senescence is described as a resistance mechanism, which can be the basis for the non-response to most common chemotherapies. It is believed that the identification of so-called senescent tumors could improve treatment strategies for solid tumors and, in particular, avoid inefficient treatment of patients with highly toxic drugs.

The aim of this study is to investigate the safety, radiation exposure (dosimetry) and diagnostic accuracy of the novel diagnostic substance [18F]FPyGal if it is used before tumor imaging imaging (here: positron emission tomography combined with magnetic resonance imaging (PET / MRT) or in combination with computed tomography (PET / CT)).

Diagnostic substances used in imaging such as [18F]FPyGal are known as radiotracers, since their distribution in the tumor tissue can provide information about the special tumor biological processes taking place there.

In the context of this study, it is of particular interest to find out whether it is possible to use the novel radiotracer [18F]FPyGal to detect areas after standard tumor therapy that contain particularly resistant (therapy-resistant) tumor cells. This resistance phenomenon in tumor tissues, which may be visualized with the radiotracer [18F]FPyGal, is called tumor senescence.

The latest research results show that senescent tumor cells can not only evade different forms of chemotherapy or radiation therapy. Senescent tumor cells can also cause the cancer to come back later. That is why current therapeutic research is concentrating on developing new approaches to combat such senescent tumor cells. For this it is relevant to be able to first diagnose senescent tumor cells as well as possible using imaging.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age at the time of signing the informed consent
* Patients with locally advanced primary non-operable solid tumors (AEGs, rectum cancers, NSCLCs, NUT midline carcinomas (NMC))
* Eastern Cooperative Oncology Group Performance (ECOG) Status ≤ 2
* Adequate bone marrow, renal, and hepatic function defined by laboratory tests within 14 days prior to study treatment:

  * Neutrophil count ≥ 1,500/mm3
  * Platelet count ≥ 100,000/µl
  * Bilirubin ≤ 1.5 x upper limit of normal (ULN)
  * ALT (alanine transaminase) and AST (aspartate transaminase) ≤ 2.5 x ULN
  * PT-INR (prothrombin time and international normalized ratio) /PTT (partial thromboplastin time)= ≤ 1.5 x ULN
  * Creatine kinase ≤ 2.5 x ULN
  * Serum creatinine ≤ 1.5 mg/dl or creatinine clearance ≥ 60 ml/min
* Patients scheduled for neo-adjuvant (radio-) chemotherapy and subsequent tumor surgery (Groups a-c) or tumor biopsy (Group d)
* Understand and voluntarily sign an informed consent document prior to any study related assessments/ procedures.
* Able to adhere to the study visit schedule and other protocol requirements
* Consent to practice double-barrier contraception until end of the study (28 days after last [18F]FPyGal injection)

  * Females of childbearing potential (FCBP) must agree

    * to use two reliable forms of contraception simultaneously or practice complete abstinence from heterosexual contact for at least 28 days before starting study drug, while participating in the study (including dose interruptions), and for at least 28 days after end of study treatment and must agree to pregnancy testing during this timeframe
    * to abstain from breastfeeding during study participation and 7 days after end of study drug administration.
  * Males must agree

    * to use a latex condom during any sexual contact with FCBP while participating in the study and for at least 28 days after end of study treatment, even if he has undergone a successful vasectomy
    * to refrain from donating semen or sperm while participating in the study and for at least 28 days after end of study treatment.

Exclusion Criteria:

* Any contraindication for MRI (impaired renal function and / or known hypersensitivity to gadolinium-containing contrast agent are not considered as contraindication, since then imaging will be performed without gadolinium contrast agent).
* Known hypersensitivity to [18F]FPyGal or its components or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product
* Administration of any kind of PET tracer within a period corresponding to 8 half-lives of the representative radionuclide (e.g. for fluorine-18: 109.77 min, 8x109.77 min =14.7 h)
* Persistent toxicity (>Grade 2) according to Common Terminology Criteria for Adverse Events [CTCAE] version 5.0, caused by previous cancer therapy, excluding alopecia
* Clinical signs of active infection (> Grade 2 according to CTCAE version 5.0)
* History of HIV infection
* Immunocompromised patients
* Active or chronic viral hepatitis (HBV or HCV)
* History of autoimmune disease
* History of relevant CNS pathology or current relevant CNS (central nervous system) pathology (e.g. seizure, paresis, aphasia, cerebrovascular ischemia/hemorrhage, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, psychosis, coordination or movement disorder) Epilepsy requiring pharmacologic treatment
* Therapeutic anticoagulation therapy
* Major surgery within 4 weeks of starting study treatment. Patients must have recovered from any effects of major surgery.
* Patients receiving any systemic chemotherapy or radio-therapy within 2 weeks prior to study treatment or a longer period depending on the defined characteristics of the agents used
* Heart failure NYHA (New York Heart Association) III/IV
* Severe obstructive or restrictive ventilation disorder
* Known history of GI-perforation
* Patients not able to declare meaningful informed consent on their own
* Women during pregnancy and lactation; female patients of childbearing potential or male patients with female partners of childbearing potential not willing to practice effective contraception by using a double-barrier method from Day 0 until 28 days post-dose.
* Male patients planning to donate sperm while participating in the study and for at least 28 days after end of study treatment.
* Participation in other clinical trials or observation period of competing trials

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | 7 days
  Incidence and severity of adverse events (AEs) (CTCAE V5.0) over 7 days Grade 1: no interruption; Grade 2: interrupt until Grade 0/1; Grade 3 and >3: interruption of study

SECONDARY OUTCOMES:
Number of patients exhibiting positive signals for senescent tumor cells in PET-imaging and/or tumor histopathology | through study completion, an average of 6 month
  Positive [18F]FPyGal-PET-imaging of patient's tumor will be correlated with histopathology using senescence specific biomarkers against SABG (senescence-associated ß-galactosidase), p16, p21, and p53

CONTACTS AND LOCATIONS:
Overall Officials: Lars Zender, MD, Study Director — University Hospital of Tübingen
Locations (1):
- University Hospital of Tübingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No